CLINICAL TRIAL: NCT04602247
Title: Evaluation of Iron Bioavailability From Iron Chlorophyllin in Young Women Using the Iron Stable Isotopic Method
Brief Title: Evaluation of Iron Bioavailability From Iron Chlorophyllin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SIC2020
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Iron Deficiency
Keywords: iron deficiency; Iron chlorophyllin
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Intervention Model Description: The study will be a single-center, prospective cross-over trial in which each subject receives all test conditions. During the screening, about 2 weeks before the start of the study, women will be assessed for eligibility. Finally, 55 eligible women will be invited to participate.
  Each subject will complete six iron absorption studies in which they will receive supplemental iron doses of 6 mg iron.The experimental phase will last for 37 days. The labeled iron doses will be administered on days 1, 3, 5, 19, 21 and 23. Since only three isotopes are used in the study, after day 5, there will be a wait period of 14 days to allow for incorporation of the labeled iron into erythrocytes. On day 19, 21 and 23 the other three test doses are administered. Randomization of the interventional products listed above will be set up as such, to ensure that participants do not receive the same isotopes in a given week. On day 1, day 19 and day 37, a venous blood sample will be collected.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- SIC (Experimental): 100 mg sodium iron chlorophyllin (SIC) containing 6 mg 57 Fe.
  Interventions: Dietary Supplement: SIC
- SIC + AA combined (Experimental): 100 mg sodium iron chlorophyllin (SIC) containing 6 mg 57 Fe given with 40 mg Ascorbic Acid
  Interventions: Dietary Supplement: SIC + AA combined
- FeSO4 (Active Comparator): 6mg of FeSO4 given as 4 mg 56Fe and 2mg 58Fe
  Interventions: Dietary Supplement: FeSO4
- FeSO4 + AA combined (Active Comparator): 6mg of FeSO4 given as 4 mg 56Fe and 2mg 58Fe along with 40 mg Ascorbic Acid
  Interventions: Dietary Supplement: FeSO4 + AA combined
- EP + FeSO4 combined (Experimental): 100 mg of Chlorophyllin without the Magnesium central atom along with 6 mg FeSO4 as 54 Fe
  Interventions: Other: EP + FeSO4 combined
- EP + FeSO4 + AA combined (Experimental): 100 mg of Chlorophyllin without the Magnesium central atom along with 6 mg FeSO4 as 54 Fe along with 40 mg of Ascorbic Acid
  Interventions: Other: EP + FeSO4 + AA combined

INTERVENTIONS:
Dietary Supplement: SIC — Sodium Iron Chlorophyllin, whose bioavailability is to be studied
  Arms: SIC
Dietary Supplement: SIC + AA combined — Sodium Iron Chlorophyllin and ascorbic acid. The ascorbic acid should not have an effect on Sodium Iron Chlorophyllin
  Arms: SIC + AA combined
Dietary Supplement: FeSO4 — Ferrous sulfate serves as a positive control, whose iron bioavailability is known
  Arms: FeSO4
Dietary Supplement: FeSO4 + AA combined — Ferrous sulfate serves as a positive control and the addition of ascorbic acid, further enhances its bioavailability
  Arms: FeSO4 + AA combined
Other: EP + FeSO4 combined — Chlorophyllin with an empty porphyrin ring, given along with FeSO4 to study if there is an incorporation of Fe into the porphyrin ring as it passes the gastric system
  Arms: EP + FeSO4 combined
Other: EP + FeSO4 + AA combined — Chlorophyllin with an empty porphyrin ring, given along with FeSO4 to study if there is an incorporation of Fe into the porphyrin ring as it passes the gastric system. Ascorbic acid is given along with the intervention to see if there is any difference in the fractional iron absorption when compared to EP+ FeSO4
  Arms: EP + FeSO4 + AA combined

SUMMARY:
The overall objective of this study is to evaluate the iron absorption from iron chlorophyllin. Iron deficiency is a public health problem in both developing and industrialized countries. There are several approaches to combat iron deficiency. Most supplements in the present day, to address the problem of iron deficiency, are in the form of iron salts, known as ferrous salts, especially ferrous sulfate. However, we can only usually absorb about 20% of the total iron content in ferrous sulfate. The common strategy of food supplement companies is to increase the amount of iron in the supplements to compensate for the low absorption rate. However, this often causes gastrointestinal side effects. In the present study, we would like to measure the iron bioavailability from sodium iron chlorophyllin, which made up from ferrous salts and chlorophyllin and where we hypothesize that it is absorbed via a different pathway than ferrous sulfate. Via this mechanism, we further hypothesize that sodium iron chlorophyllin will therefore have an enhanced bioavailability and more favorable side effect profile than ferrous sulfate and other iron salts.

DETAILED DESCRIPTION:
New approaches to treat iron deficiency include developing novel iron compounds with possible iron absorption routes that increase iron bioavailability and reduce gastrointestinal side effects. Heme iron is considered to be highly bioavailable (10-20%) and less affected by meal composition than non-heme iron. Heme iron is iron (Fe2+) that is bound to the iron protoporphyrin IX prosthetic groups of proteins, mainly hemoglobin and myoglobin, which are present in animal tissue. Heme is released from hemoglobin during digestion so that it can be taken up by the duodenal enterocytes. The intact iron porphyrin is transported across the brush border membrane by the Heme Carrier Protein 1 (HCP1). Once inside the cell, the iron is released, and it is then likely to enter the low molecular weight pool of iron. The use of heme analogues from vegetable origin could provide an alternative iron source of potentially high bioavailability.

Sodium iron chlorophyllin (SIC) is a water-soluble semisynthetic chlorophyll derivative where the magnesium in the porphyrin ring has been substituted by iron. It is a greenish brown pigment that dissolves in water, alcohols, and chloroform, but not ethers. SIC is known to have a superior processing stability to chlorophyll and is commonly used as food colorings in Asian countries including in Korea and Japan, for foods that do not contain meat or fish. Magnesium Chlorophyllin has an E number of E140 and is approved as a food additive in Europe. Currently sodium iron chlorophyllin is present in the Designated Additives List in Japan with a number 261. Designated additives are those designated by the Minister of Health, Labour and Welfare as substances that are unlikely to harm human health based on Article 10 of the Food Sanitation Act.

Given the porphyrin ring heme-like structure of SIC, it may be an alternative delivery route for iron, suitable also for vegetarians and vegans, yet there are few studies investigating the use of SIC for this purpose.

A recent study by Ding et al. 2019 suggests a positive effect of SIC on hemoglobin (Hb) values in iron-deficiency anemia (IDA) in children and adults after 1 month of treatment. They assume that SIC is taken up by the heme carrier protein. The researchers used shengxuening tablets, also known as SXN, which are based on chlorophyll/porphyrin structures extracted from silkworms in which the Mg is replaced by the Fe and then coadjutants are added. This study provided no data on the absorption pathway of the SXN compound. Thus, it remains unclear if it was taken up by the heme transporter or whether it was digested and the Fe released in the gut lumen to join the non heme Fe pool, and thereby improved Hb in the IDA subjects. The authors also describe Xray diffraction assays to assess if the chlorophyllin porphyrin ring contained Fe and not Mg, however these data are not reported.

Miret et al. (2010) studied the stability of heme-analogous SIC absorption using the Caco-2 cell model. The SIC remained stable and only 5% of the Fe from the compound was released at pH 2 to 4. In-house dissolution studies conducted at the Human Nutrition Laboratory (HNL) show only a 2% release of Fe from the compound at similar pH levels. Using solid phase extraction at a higher pH of 7, similar to that in the duodenum, we observed a 5% Fe loss, which may correspond to free iron or iron liberated from any other binding sites on the chlorophyll structure.

Toyoda et al. (2014) performed a toxicity study of SIC performed in male and female rats with oral administration of SIC in their diet at concentrations of 0%, 0.2%, 1.0%, and 5.0% for 13 weeks. No abnormal clinical signs, no mortality and no abnormal hematological changes were observed in any of the groups during the experiment. Based on the histopathology of the parotid glands, the no-observed-adverse-effect level (NOAEL) of SIC in this study was estimated to be 1.0% (609 mg SIC/kg bodyweight (bw)/day for males and 678 mg/kg bw/day for females). In the present study, we will use 6 mg elemental iron, in 100 mg SIC, 0.002% of the equivalent dose administered by Toyoda et al.

SIC has been produced at the HNL with a 75% incorporation of iron into the chlorophyll. Our protocol is based on a Unilever patent that is no longer active, with in-house adaptation. The SIC has a neutral taste and will be presented as a dark green liquid, being the solution of SIC in water.

The goal of this project is to develop a novel iron compound that can be used as a food supplement. The iron content in our SIC will be limited to 6 mg per dose, which therefore does not exceed the 14 mg daily iron dose stipulated as the legal maximum in Switzerland for food supplements. SIC is already used widely as a food colorant and is safe for human consumption.

We propose to test our SIC against a known comparator, ferrous sulfate, to ascertain whether SIC is an effective iron delivery compound. If SIC, as hypothesized, behaves in a similar way to heme, then commonly used enhancers of iron absorption effective on ferrous sulfate, such as ascorbic acid, will not have an effect on the absorption of iron from SIC

ELIGIBILITY:
Inclusion Criteria:

* female aged between 18-45 y old;
* SF <80 µg/L;
* BMI 18.5-24.9 kg/m2;
* weight <70 kg;
* signed informed consent;
* able to communicate and comprehend English language

Exclusion Criteria:

* anemia (Hb <12 g/dL);
* inflammation (CRP > 5 mg/L);
* chronic digestive, renal and/or metabolic disease;
* chronic medications (except for oral contraceptives);
* use of vitamin, mineral and pre- and/or probiotic supplements in the previous 2 weeks before study initiation and during the course of the study;
* blood transfusion, blood donation or significant blood loss over the past 4 months;
* pregnancy (tested in serum at screening) or intention to become pregnant;
* lactation up to 6 weeks before study initiation;
* earlier participation in a study using stable isotopes or participation in any clinical study within the last 30 days;
* smoking;
* unwilling to use an effective method of contraception.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 55 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Fractional Iron Absorption | day 19
  Fractional iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of the intervention products .Fractional iron absorption will be measured as erythrocyte incorporation of the naturally occurring iron forms with different masses used to label the iron supplements.
Fractional Iron Absorption | day 37
  Fractional iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of the intervention products .Fractional iron absorption will be measured as erythrocyte incorporation of the naturally occurring iron forms with different masses used to label the iron supplements.

SECONDARY OUTCOMES:
Hemoglobin | Day 1, day 19 and day 37 of the study
  Iron status marker
Plasma Ferritin | Day 1, day 19 and day 37 of the study
  Iron status marker
soluble transferrin receptor (sTfR) | Day 1, day 19 and day 37 of the study
  Iron status marker
C-Reactive Protein | Day 1, day 19 and day 37 of the study
  Inflammation marker

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Zürich, Laboratory of Human Nutrition, Zurich, Canton of Zurich, Switzerland